CLINICAL TRIAL: NCT05516147
Title: SAFE at Home: A Service to Provide Social Engagement to Community-Dwelling Persons With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopeful Aging (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R43AG075974 (NIH)
Record Dates: First submitted 2022-08-10; First posted 2022-08-25 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer Disease; Dementia; Dementia, Vascular; Dementia, Mixed
Keywords: non-pharmacological intervention; psychosocial
MeSH Terms: conditions — Alzheimer Disease; Dementia; Dementia, Vascular; Mixed Dementias

STUDY DESIGN:
Intervention Model Description: All participants receive the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): SAFE at Home Intervention
  Interventions: Behavioral: SAFE at Home

INTERVENTIONS:
Behavioral: SAFE at Home — SAFE at Home will enable community-dwelling PWD to participate in videoconference-based group activities with their peers, that is, other PWD. SaH sessions will be facilitated by highly trained Engagement Professionals.

SUMMARY:
The proposed Phase 1 study will involve initial development and evaluation of a new service called Social Activities For Engagement at Home or SAFE at Home (SaH). SaH will enable PWD to participate in videoconference-based group activities with their peers-i.e., other PWD. SaH sessions will be facilitated by highly trained "Engagement Professionals," who will be SaH staff members that have a background in recreation therapy, activity coordination, or a similar field. The proposed study has three Specific Aims: Aim 1. Develop an Alpha version of the SaH app, including app infrastructure and preliminary activity content for live group sessions, as well as staff training and coaching modules. Aim 2. Examine the app's acceptability/feasibility (by assessing attendance, session length, and engagement/affect). Aim 3. Examine satisfaction with the app by directly eliciting feedback from PWD and life enrichment staff.

DETAILED DESCRIPTION:
Aim 1. Develop an Alpha version of the SAFE at Home app, including app infrastructure and preliminary activity content for live group sessions, as well as staff training and coaching modules. During Months 1-6, the Development Team (DT) will create the initial product design and prototype for use in the study. The study team will engage 5 PWD, 5 family members, and 5 activity professionals in focus groups to review the mockups and to understand end user preferences in terms of user experience and activity content. This will be the only involvement for these participants. New participants will be recruited for the quasi-experiment (described below). Aim 2. Examine the app's acceptability/feasibility (by assessing attendance, session length, and engagement/affect) During Months 5-10, the Experimental Team (ET) will utilize a quasi-experimental pre-post design (i.e., baseline vs. treatment / post-treatment) to conduct a two-month long acceptability and feasibility trial of SaH. During this trial 15 PWD, 15 Family Members, and 5 Life Enrichment professionals will use the product to determine functionality, acceptability, and feasibility. Baseline and Onboarding (Month 7). PWD: During the 4-week baseline period, the ET will collect the following data. PWD Demographics, medications, diagnoses, and type of dementia will be collected via proxy (family member) interview. The following assessments will be administered directly: the Short Portable Mental Status Questionnaire (SPMSQ-T), the Dementia Quality of Life Scale (DEMQOL), the Geriatric Depression Scale-Short Form (GDS-SF), and the UCLA Loneliness Scale (ULS). Researchers will interview family members (FMs) using the Neuropsychiatric Inventory-Nursing Home (NPI-NH). Using the Menorah Park Engagement Scale. researchers will observe PWD engagement and affect via videoconference on four days. This will allow us to determine "normal/baseline" engagement levels for each PWD and serve as a comparison for SaH. At the conclusion of the Baseline data collection, the ET will use the Get to Know You Portal with each PWD to determine their Cognitive and Communication levels as well as their interests. For the purposes of testing the feasibility of the SaH intervention, all group assignments will be made solely through the use of SaH tools. Staff Demographics will be collected. Staff will also take pre-training quizzes prior to taking the training modules. Family Members (FMs) will provide demographic information and serve as proxies for the above PWD measures. Intervention Period (Months 8-9). PWD: During the 8-week intervention period, PWD will participate in SaH sessions through the Social Engagement Portal. Sessions will occur twice per week and last 30-45 minutes. Staff: Staff will take the training modules developed in Aim 1 and will also run a simulated group and provide feedback. FMs will be involved simply by helping set up the hardware and helping their loved one with technical issues as needed (e.g., reconnecting to the videoconference if the connection is lost). Post Intervention Period (Month 10). PWD: The DEMQOL, GDS-SF, ULS, and NPI-NH will be re-administered at Post-Intervention, allowing us to investigate possible long-term effects. Changes on these longer-term measures are not expected in this Phase 1 study. However, data will be used to conduct power analyses for Phase 2. Staff: Staff will take post-training quizzes after completing the training modules. FMs will serve as proxies for some of the above measures. Milestones. This Aim will be considered successfully met if: (1) At least 85% of PWD agree to take part in 80% of the sessions. (2) Mean session length is least 25 minutes. (3) PWD exhibit higher levels of positive engagement/affect and lower levels of negative engagement during SaH sessions, as compared to baseline (based upon the MPES). This will be assessed by using paired samples t-tests. With the proposed sample, there will be a power of 99% to detect effects. A detailed power analysis is included in Clinical Trials-Statistical Design and Power. (4) Staff show an increase in knowledge after taking the training modules, based upon paired samples t-tests (pre-training quizzes vs. post-training quizzes). Aim 3. Examine satisfaction with the app by directly eliciting feedback from PWD and life enrichment staff. Overview: This Aim occurs concurrently with the Intervention Period for Aim 2 and utilizes the same sample and procedures-it merely tracks separate outcomes. Intervention Period (Months 8-9). PWD: During the intervention period, PWD will answer questions related to satisfaction at the end of each session. Staff: Staff will answer satisfaction questions related to the course and to the app (after the run a simulated group). FMs will answer satisfaction questions at the end of the study. Challenges. Since this aim occurs concurrently with Aim 2, no distinct challenges related solely to Aim 3 are expected. Milestones: This Aim will be considered successfully met if PWD, staff members, and FMs report high satisfaction with the app, defined as 85% being satisfied or very satisfied.

ELIGIBILITY:
PWD Inclusion Criteria:

* 65+ years old
* speak and read conversational English
* diagnosed with dementia (any type)

PWD Exclusion Criteria:

-signs of rapid cognitive decline or physical deterioration over the last six months, as evidenced by medical records.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-01-19 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Skrajner, MA, Principal Investigator — The Hearthstone Institute
Locations (1):
- Hopeful Aging, Winchester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 10
Completed | 8
Not Completed | 2
Not completed — Scheduling Conflicts Made it Impossible for them to participate | 2

BASELINE CHARACTERISTICS:
Population: All participants who enrolled, including those who could not complete due to scheduling conflicts
Arm/Group | Treatment
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 82.40 (5.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Constructive Engagement Mean on Menorah Park Engagement Scale
Description: Constructive Engagement on the Menorah Park Engagement Scale (MPES) is defined as doing or commenting on something related to the target activity. For each participant, multiple BRAIN activities were observed during weeks 5-10. Based upon all of these observations that occured during this time period, a single mean score was calculated for each participant on this MPES item. The minimum value for Constructive Engagement is zero (0) and the maximum score is two (2). Higher scores represent a better outcome. A one-sample t-test was used to assess whether the mean was different from a known Constructive Engagement mean of 0.85 for standard programming.
Time Frame: Treatment (Weeks 5-10)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 10
score on a scale | 1.22 (0.32)
Statistical Analysis 1: Comparison: Treatment; A one-sample t-test was used to assess whether the mean was different from a known Constructive Engagement mean of 0.85 for standard programming; Test type: Superiority; p < .01, t-test, 2 sided — A one-sample t-test was used to assess whether the mean was different from a known Constructive Engagement mean of 0.85 for standard programming

2. Primary Outcome: Passive Engagement Mean on Menorah Park Engagement Scale
Description: Passive Engagement on the Menorah Park Engagement Scale is defined as listening or watching something related to the target activity. For each participant, multiple BRAIN activities were observed during weeks 5-10. Based upon all of these observations that occured during this time period, a single mean score was calculated for each participant on this MPES item. The minimum value for Passive Engagement is zero (0) and the maximum score is two (2). Higher scores represent a better outcome. A one-sample t-test was used to assess whether the mean was different from a known Passive Engagement mean of 1.06 for standard programming.
Time Frame: Treatment (Weeks 5-10)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 10
score on a scale | 1.65 (0.25)
Statistical Analysis 1: Comparison: Treatment; A one-sample t-test was used to assess whether the mean was different from a known Passive Engagement mean of 1.06 for standard programming; Test type: Superiority; p < .01, t-test, 2 sided — A one-sample t-test was used to assess whether the mean was different from a known Passive Engagement mean of 1.06 for standard programming; A one-sample t-test was used to assess whether the mean was different from a known Passive Engagement mean of 1.06 for standard programming

3. Primary Outcome: Other Engagement Mean on Menorah Park Engagement Scale
Description: Other Engagement on the Menorah Park Engagement Scale is defined as doing, commenting, listening, or watching something NOT related to the target activity. For each participant, multiple BRAIN activities were observed during weeks 5-10. Based upon all of these observations that occured during this time period, a single mean score was calculated for each participant on this MPES item. The minimum value for Other Engagement is zero (0) and the maximum score is two (2). Lower scores represent a better outcome. A one-sample t-test was used to assess whether the mean was different from a known Other Engagement mean of 0.42 for standard programming.
Time Frame: Treatment (Weeks 5-10)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 10
score on a scale | 0.17 (0.36)
Statistical Analysis 1: Comparison: Treatment; A one-sample t-test was used to assess whether the mean was different from a known Other Engagement mean of 0.42 for standard programming; Test type: Superiority; p = 0.06, t-test, 2 sided — A one-sample t-test was used to assess whether the mean was different from a known Other Engagement mean of 0.42 for standard programming; A one-sample t-test was used to assess whether the mean was different from a known Other Engagement mean of 0.42 for standard programming

4. Primary Outcome: Non Engagement Mean on Menorah Park Engagement Scale
Description: Non-Engagement on the Menorah Park Engagement Scale is defined as sleeping and/or staring into space. For each participant, multiple BRAIN activities were observed during weeks 5-10. Based upon all of these observations that occured during this time period, a single mean score was calculated for each participant on this MPES item. The minimum value for Non Engagement is zero (0) and the maximum score is two (2). Lower scores represent a better outcome. A one-sample t-test was used to assess whether the mean was different from a known Non Engagement mean of 0.40 for standard programming.
Time Frame: Treatment (Weeks 5-10)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 10
score on a scale | 0.001 (0.003)
Statistical Analysis 1: Comparison: Treatment; A one-sample t-test was used to assess whether the mean was different from a known Non Engagement mean of 0.40 for standard programming; Test type: Superiority; p < .01, t-test, 2 sided

5. Primary Outcome: Pleasure Mean on Menorah Park Engagement Scale
Description: Pleasure on the Menorah Park Engagement Scale is defined as clearly observable laughing or smiling.For each participant, multiple BRAIN activities were observed during weeks 5-10. Based upon all of these observations that occured during this time period, a single mean score was calculated for each participant on this MPES item. The minimum value for Non Engagement is zero (0) and the maximum score is two (2). Lower scores represent a better outcome. A one-sample t-test was used to assess whether the mean was different from a known Non Engagement mean of 0.28 for standard programming.
Time Frame: Treatment (Weeks 5-10)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 10
score on a scale | 0.72 (0.27)

6. Secondary Outcome: Change From Baseline to Treatment on Dementia Related Quality of Life (DEMQOL)
Description: The Dementia Related Quality of Life Scale is a 28 item scale that examines quality of life in persons with dementia. The score ranges for 28 to 112. Higher scores represent a better outcome.
Time Frame: Baseline (Weeks 1-4) and Post-Treatment (Week 11)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 8
score on a scale | 0.85 (9.4)
Statistical Analysis 1: Comparison: Treatment; baseline score vs. post-treatment, paired sample t-test; Test type: Superiority; p = 0.81, t-test, 2 sided

7. Secondary Outcome: Change From Baseline to Treatment on the Neuropsychiatric Inventory-Nursing Home (NPI-NH), Frequency x Severity Score (FxS)
Description: The NPI-NH examines 10 types of neuropsychiatric symptoms in persons with dementia, with the FxS score looking creating a composite score that takes into account frequency and severity of the symtoms. The score ranges from 0 to 120. Lower scores represent a better outcome.
Time Frame: Baseline (Weeks 1-4) and Post-Treatment (Week 11)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 8
score on a scale | -3.38 (6.68)
Statistical Analysis 1: Comparison: Treatment; baseline vs. post-treatment, paired sample t-test; Test type: Superiority; p = 0.20, t-test, 2 sided

8. Secondary Outcome: Change From Baseline to Treatment on the University of California, Los Angels (UCLA) Loneliness Scale
Description: The UCLA Loneliness Scale is a widely used psychological tool designed to measure an individual's subjective feelings of loneliness and social isolation. The 20-item version consists of statements related to social connections, with responses typically rated on a four-point Likert scale (e.g., "Never," "Rarely," "Sometimes," "Often"). Scoring involves summing item responses, with higher scores indicating greater levels of loneliness. The range of total possible score is 20 (least amount of loneliness) to 80 (most amount of loneliness).
Time Frame: Baseline (Weeks 1-4) and Post-Treatment (Week 11)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 8
score on a scale | -0.71 (8.94)
Statistical Analysis 1: Comparison: Treatment; baseline vs. post-treatment, paired sample t-test; Test type: Superiority; p = 0.83, t-test, 2 sided

9. Secondary Outcome: Change From Baseline to Treatment on the Geriatric Depression Scale-Short Form (GDS-SF)
Description: The 15-item Geriatric Depression Scale (GDS-SF) is a screening tool used to assess depressive symptoms in older adults. Each item is answered with a "Yes" or "No"** response, with a total score ranging from 0 to 15, where higher scores indicate greater depressive symptoms. A score of 5 or more** suggests possible depression, warranting further clinical evaluation.
Time Frame: Baseline (Weeks 1-4) and Post-Treatment (Week 11)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 8
score on a scale | -1.00 (2.67)
Statistical Analysis 1: Comparison: Treatment; baseline vs. post-treatment, paired sample t-test; Test type: Superiority; p = 0.320, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 2.5 months
Description: Participants and/or family members of participants were asked to let the Principal Investigator (PI) know (via email, phone, or in person) about adverse events if/when they occur. In addition, each site was contacted via email at the end of each month by the PI. In that email, the PI asked the long-term care community whether any adverse events had occurred that had not yet been reported.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-12-01): https://cdn.clinicaltrials.gov/large-docs/47/NCT05516147/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-01): https://cdn.clinicaltrials.gov/large-docs/47/NCT05516147/SAP_001.pdf